CLINICAL TRIAL: NCT03041597
Title: An Randomized Controlled Trial Comparing Immediate Loading With Conventional Loading Using Cone-anchored Implant Supported Removable Dental Prostheses, a Two Year Follow up
Brief Title: Dental Implant Supported Removable Dental Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Lauren Bernard, Periodontist, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B32220096198
Record Dates: First submitted 2017-01-26; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Implant Complication; Prosthesis Survival
MeSH Terms: conditions — Prosthesis Failure | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate loading (Experimental)
  Interventions: Procedure: placement of implants; Procedure: immediate loading; Device: Ankylos implant
- delayed loading (Active Comparator)
  Interventions: Procedure: placement of implants; Procedure: conventional loading; Device: Ankylos implant

INTERVENTIONS:
Procedure: placement of implants — surgical procedure and placement of implants
Procedure: immediate loading — cone-anchored implant supported removable dental prostheses placement
  Arms: Immediate loading
Procedure: conventional loading — cone-anchored implant supported removable dental prostheses placement in 3mo
  Arms: delayed loading
Device: Ankylos implant

SUMMARY:
To prospectively monitor the survival rate of Ankylos® dental implants, comparing delayed versus immediate loading, using abutments with the SynCone® concept for implant-supported detachable dental prosthesis (ISDDP) in the edentulous upper jaw.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Extraction sockets should have healed at least 4 months
* Sufficient bone volume to place six implants in the maxilla
* No previous bone augmentation procedures
* The mandible can have any kind of dentition as long as a well-distributed contact relationship with the new prosthesis in the maxilla can be established.
* Accepting to comply with study procedures

Exclusion Criteria:

* Physical or psychological disorders prohibiting implant treatment
* Heavy smoking (>10 cigarettes/day)
* Present alcohol and/or drug abuse
* Physical handicap that may interfere with the ability to perform oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
bone loss | Difference between loading and Year two
  measured in mm op peri-apical radiography. Mesial and Distal measurement of implant.

SECONDARY OUTCOMES:
probing pocket depth | Difference between loading and Year two
  Measurement in mm, 4 sites per implant.
plaque | Difference between loading and Year two
  presence of plaque, 4 sites per implant, Yes=1 or No=0
bleeding on probing | Difference between loading and Year two
  presence of bleeding on probing, 4 sites per implant, Yes=1 or No=0

IPD SHARING:
Plan to Share IPD: Undecided